CLINICAL TRIAL: NCT06257342
Title: Physical Abilities of Teenagers With Familial Mediterranean Fever
Acronym: Sport & FMF
Status: Active, not recruiting | Type: Observational
Sponsor: Véronique Hentgen (Other)
Responsible Party: Sponsor-Investigator, Véronique Hentgen, Professor, Versailles Hospital
Organization: Versailles Hospital (Other)
Other Study IDs: P23/04
Record Dates: First submitted 2024-02-06; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-06

CONDITIONS: Familial Mediterranean Fever
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — Walking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: 6 minutes walk — A 6 minutes walk test

SUMMARY:
Physical abilities of teenagers with familial Mediterranean fever

DETAILED DESCRIPTION:
Physical abilities of teenagers with familial Mediterranean fever by describing the maximum oxygen consumption (VO2max) estimated from a 6-minute walk test

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of FMF according to the Tel-Hashomer criteria for whom a sports evaluation was offered during their bridging program
* Age >12
* Followed or having been followed in the pediatric department of the CH of Versailles
* No opposition of the patient and his/her parent/legal guardian in case of a minor patient

Exclusion Criteria:

Expressed refusal of the patient and his/her parent/legal guardian to participate in the study and/or to use genetic data for research purposes

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Teenagers with familian mediteranean fever
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-07-30 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the maximum oxygen consumption (VO2max) estimated from the 6-minute walk test | 6 minutes
  Describe the maximum oxygen consumption (VO2max) estimated from the 6-minute walk test

CONTACTS AND LOCATIONS:
Locations (1):
- CH de Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No